CLINICAL TRIAL: NCT00471224
Title: A Prospective Safety Follow Up Study Of Subjects Enrolled In Study A4321001 And Who Have Received Formulated Drug Product (LOT 8716-098).
Brief Title: A Prospective Safety Follow Up Study Of Subjects Enrolled In Study A4321001 And Who Have Received Drug Product
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Other Study IDs: A4321004
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Siderosis
MeSH Terms: conditions — Siderosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who have received drug.: Patients who have received drug.
  Interventions: Other: Observational Trial

INTERVENTIONS:
Other: Observational Trial — No intervention is being used in this study.

SUMMARY:
This protocol intends to detail investigations necessary to evaluate the ocular safety of subjects enrolled in study A4321001 and who have received formulated Drug Product (Lot 8716-098).

ELIGIBILITY:
Inclusion Criteria:

* A subset of subjects enrolled in study A4321001 and who have received formulated drug product (Lot 8716-098) will be included in the safety follow up study.

Exclusion Criteria:

None

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A subset of subjects enrolled in study A4321001 and who have received formulated drug product.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
follow up for ocular safety and clinical features of ocular siderosis | 12 months

SECONDARY OUTCOMES:
ERG changes | 12 months
Anterior segment and fundal photography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4321004&StudyName=A%20Prospective%20Safety%20Follow%20Up%20Study%20Of%20Subjects%20Enrolled%20In%20Study%20A4321001%20And%20Who%20Have%20Received%20Drug%20Product